CLINICAL TRIAL: NCT02359734
Title: A National Study of Intravenous Medication Errors: Understanding How to Improve Intravenous Safety With Smart Pumps
Brief Title: A National Study of Intravenous Medication Errors
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Johns Hopkins University (Other); Winchester Medical Center (Other); Central DuPage Hospital (Other); Vanderbilt University (Other); Massachusetts General Hospital (Other); University of California, San Diego (Other); Valleywise Health (Other); Danbury Hospital (Other); Association for the Advancement of Medical Instrumentation (Other); CareFusion foundation (Unknown); Candler Hospital (Unknown)
Responsible Party: Principal Investigator, David W. Bates, MD, MSc, Chief, Division of General Medicine, Brigham and Women's Hospital
Other Study IDs: 2012P000709
Record Dates: First submitted 2015-01-05; First posted 2015-02-10 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Medication Administered in Error
Keywords: Patient safety; Medication errors; Smart infusion pump

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Brigham and Women's Hospital.: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Brigham and Women's Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Johns Hopkins University Hospital: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Johns Hopkins University Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Winchester Medical Center: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Winchester Medical Center. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Central DuPage Hospital: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Central DuPage Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Vanderbilt University: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Vanderbilt University Medical Center. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Massachusetts General Hospital: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Massachusetts General Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- University of California, San Diego: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at University of California, San Diego. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Maricopa Integrated Health System: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Maricopa Integrated Health System. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Danbury Hospital: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Danbury Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump
- Candler Hospital: Patients who had IV medications with smart pumps in one surgical unit, one medical unit, one Medical ICU, and one surgical ICU at Candler Hospital. In these unit, the intervention bundle was implemented.
  Interventions: Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump

INTERVENTIONS:
Other: Smart pump safety Intervention bundle for improving IV medication administration process with smart pump — Smart pump safety intervention bundle includes three components--1) eliminating unauthorized medications; implement standardized discontinuation policy of medications, implement standardized keep vein open rates and keep vein open rate order sets, and implement standardized verbal order practice. 2) Implement standardized intravenous(IV) labeling and IV tubing labels. 3) Implement standardized drug library lists and drug library use policies

SUMMARY:
To identify the key issues around use of computerized patient infusion devices (called "smart pumps").

To develop strategies that will improve the prevention of intravenous errors that will be broadly applicable.

The investigators will conduct a national study using the general methodology developed by Husch et al. to allow a rapid assessment of the frequency and types of medication errors at an institution.

The key questions the investigators will address are:

1. What are the frequency and types of intravenous medication errors?
2. How much variability is there by frequency and type among settings?
3. After review of the initial data, what strategies appear to have the greatest potential for reducing intravenous medication error frequency?
4. How effective is an intervention including a bundle of these strategies at multiple sites?

DETAILED DESCRIPTION:
Overall Study Design: This is a multi-hospital study to investigate medication errors using smart pumps. The proposed study will be conducted over three phases for a total of 36 months phases. In Year 1, an observational study will be conducted by investigators at ten multiple hospital sites. The investigators will prospectively compare the medication, dose, and infusion rate on the IV pump with the prescribed medication, doses, and rate in the medical record. Preventability with smart pump technology will be retrospectively determined based on a rigorous definition of currently available technology. The investigators will also make comparisons across sites by overall rate and degree of variability among sites.

Then, in Year 2, these results will be evaluated, and a consensus process including a face-to-face meeting will take place to evaluate the types of events and to develop an intervention which will be implemented at multiple sites. After a run-in period, the intervention will be tested in Year 3 at the sites, and the data will be analyzed, and the investigators will produce a report and a set of recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients if they receive any IV fluid or medication on the day of observation in the study units.

Exclusion Criteria:

* patients who are under 21 years old.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Any patients who are hospitalized in Medical ICU, surgical ICU, medicine unit and surgical unit on the day of data collection
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incident rates of wrong dose | Two years
  The same medication but the dose is different from the prescribed order.
Incident rates of wrong rate | Two years
  A different rate is displayed on the pump from that prescribed in the medical record. Also refers to weight based doses calculated incorrectly including using a wrong weight.
Incident rates of wrong concentration | Two years
  An amount of a medication in a unit of solution that is different from the prescribed order.
Incident rates of wrong IV fluids/medications | Two years
  A different fluid/medication as documented on the IV bag label is being infused compared with the order in the medical record.
Incident rates of delay of medication administration | Two years
  An order to start or change medication or rate not carried out within 4 hours of the written order or intended start time per institution policy.
Incident rates of omission of IV fluids/medications | Two years
  The medication ordered was not administered to a patient or administered anytime after 4 hours of the intended start time.
Incident rates of unauthorized medication | Two years
  Fluids/medications are administered to the patient but no order is present in medical record. This includes failure to document a verbal order.
Incident rates of patient identification (ID) error (wrong patient) | Two years
  Patient either has no ID band on or information on the ID band or label is incorrect.
Incident rates of smart pump or drug library not used | Two years
  Smart pump is not used (bypassing smart pump) or smart pump was used but the drug library was not selected, rather manual entry mode was used (bypassing drug library)
Incident rates of oversight allergy | Two years
  Medication is administered to a patient with a known allergy to the drug or class.
Incident rates of pump setting error | Two years
  Setting programmed into the pump is different from the prescribed order.
Compliance rate of label not complete according to policy | Two years
  Documented information on the medication label is different from required information per institution policy.
Compliance rate of IV tubing not tagged according to policy | Two years
  IV tubing change label is not tagged per institution policy.
Incident rates of expired drug | Two years
  The expiration date or time of the fluids/medications has passed.
Overall medication errors | Two years
  Total number of all observed medication errors(including outcome 1-14)
Higher-severity medication errors | Two years
  All medication errors with an NCC MERP severity rating of C or greater (excluding violation of hospital policy errors;outcome 12 and 13).

SECONDARY OUTCOMES:
Compliance rate of using smart pump use | Two years
  Compliance rate of using smart pump
Compliance rate of using drug library use | Two years
  Compliance rate of using drug library
Potential adverse drug events | Two years
  Medication errors with potential for harm categorized as D (errors that would have required increased monitoring to preclude harm) or higher by NCC MERP Index

CONTACTS AND LOCATIONS:
Overall Officials: David W Bates, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Schnock KO, Dykes PC, Albert J, Ariosto D, Call R, Cameron C, Carroll DL, Drucker AG, Fang L, Garcia-Palm CA, Husch MM, Maddox RR, McDonald N, McGuire J, Rafie S, Robertson E, Saine D, Sawyer MD, Smith LP, Stinger KD, Vanderveen TW, Wade E, Yoon CS, Lipsitz S, Bates DW. The frequency of intravenous medication administration errors related to smart infusion pumps: a multihospital observational study. BMJ Qual Saf. 2017 Feb;26(2):131-140. doi: 10.1136/bmjqs-2015-004465. Epub 2016 Feb 23. PMID 26908900
- [Derived] Schnock KO, Dykes PC, Albert J, Ariosto D, Cameron C, Carroll DL, Donahue M, Drucker AG, Duncan R, Fang L, Husch M, McDonald N, Maddox RR, McGuire J, Rafie S, Robertson E, Sawyer M, Wade E, Yoon CS, Lipsitz S, Bates DW. A Multi-hospital Before-After Observational Study Using a Point-Prevalence Approach with an Infusion Safety Intervention Bundle to Reduce Intravenous Medication Administration Errors. Drug Saf. 2018 Jun;41(6):591-602. doi: 10.1007/s40264-018-0637-3. PMID 29411338